CLINICAL TRIAL: NCT04614168
Title: Can Maximising Time in Range Using Automated Insulin Delivery and a Low Carbohydrate Diet Restore the Glucagon Response to Hypoglycaemic in Type 1 Diabetes?
Brief Title: Maximising Time With a Normal Blood Glucose to Restore the Glucagon Response in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); The Leona M. and Harry B. Helmsley Charitable Trust (Other); Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AC19163
Record Dates: First submitted 2020-10-07; First posted 2020-11-03 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes; Type 1 Diabetes Mellitus With Hypoglycemia; Hypoglycemia; Hypoglycemia Unawareness; Glucagon Deficiency; Insulin Hypoglycemia
Keywords: Type 1 diabetes; Hypoglycaemia; Hypoglycemia; Glucagon; Insulin; Low carbohydrate diet; Stable isotope
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Insulin Infusion Systems; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups using stratified sampling to match for age, sex and BMI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 - Standard Care (Active Comparator): This group will continue on their standard diabetes care. They will be required to undergo three periods of blinded continuous glucose monitoring each lasting 20-days at: baseline, 4 months and 8 months. Participants in this group will undergo a hyperinsulinaemic hypoglycaemic clamp study at baseline and 8 months. They will also complete quality of life and diabetes treatment questionnaires at baseline and 8 months.
  Interventions: Procedure: Stepped hyperinsulinaemic-hypoglycaemic clamp study; Device: Blinded continuous glucose monitor; Procedure: Stable isotope studies- D2 Glucose and D5 Glycerol
- Group 2- Automated insulin delivery and low carbohydrate diet (Experimental): This group will be placed on an automated insulin delivery system: Tandem t:slim x2 insulin pump with Control IQ technology and Dexcom G6 continuous glucose monitor. They will also be asked to follow a low-carbohydrate diet of 30-40g of carbohydrate per main meal. At baseline they will have a 20-day period of blinded continuous glucose monitoring. Participants in this group will undergo a stepped hyperinsulinaemic hypoglycaemic clamp study at baseline and 8 months. They will also complete quality of life and diabetes treatment questionnaires at baseline and 8 months.
  Interventions: Procedure: Stepped hyperinsulinaemic-hypoglycaemic clamp study; Device: Insulin pump; Device: Continuous glucose monitor; Other: Low carbohydrate diet; Device: Blinded continuous glucose monitor; Procedure: Stable isotope studies- D2 Glucose and D5 Glycerol

INTERVENTIONS:
Procedure: Stepped hyperinsulinaemic-hypoglycaemic clamp study — Participants will commence on a primed insulin infusion at a constant rate of 60mU/m2/min along with a variable rate 20% glucose infusion. Participants will have their blood glucose monitored every 5 minutes. The glucose infusion will be altered to achieve the desired blood glucose plateaus of: 5mmol/l, 3mmol/l and 2.5mmol/l. Each plateau will be held for 40 minutes. During each plateau blood samples will be taken on three occasions for: glucagon, cortisol, adrenaline, noradrenaline, D2 glucose and D5 glycerol. On two occasions during each plateau participants will complete the Edinburgh hypoglycaemia scale and the following cognitive tests: trail making test, digit span test, digit symbol substitution test and four choice reaction time test. At the end of the clamp study the insulin infusion will be discontinued and the blood glucose will be allowed to rise to the normal range. Participants will consume lunch before leaving the clinical research facility.
Device: Insulin pump — Insulin pump with a built-in algorithm that allows it to work with a CGM device to adjust insulin delivery based on CGM readings.
  Other Names: Tandem t:slim x2 with Control IQ technology
  Arms: Group 2- Automated insulin delivery and low carbohydrate diet
Device: Continuous glucose monitor — Continuous glucose monitoring device that sends data to the insulin pump to allow the algorithm to adjust insulin delivery. Participants are able to see the glucose data from the device when it is used in open mode.
  Other Names: Dexcom G6
  Arms: Group 2- Automated insulin delivery and low carbohydrate diet
Other: Low carbohydrate diet — 30-40g of carbohydrate per main meal portion.
  Arms: Group 2- Automated insulin delivery and low carbohydrate diet
Device: Blinded continuous glucose monitor — Allows data on blood glucose to be collected without values altering the behaviour of the participant. Participants have to continue to monitor their own blood glucose while wearing the device in the blinded mode.
  Other Names: Dexcom G6
Procedure: Stable isotope studies- D2 Glucose and D5 Glycerol — These studies will take place at the same time as the hyperinsulinaemic hypoglycaemic clamp studies. Participants will receive a priming dose of each stable isotope followed by a continuous infusion for the remainder of the clamp study.

SUMMARY:
Almost all people who have had type 1 diabetes for 5 years have a defect in secretion of the hormone Glucagon. This hormone is involved in the body's response to low blood glucose (hypoglycaemia). It works by releasing glucose stores from the liver to bring the blood glucose back to normal. This defect therefore increases the risk of severe hypoglycaemia. The reason for this Glucagon defect in people with Type 1 diabetes is currently unknown.

This study aims to look at the Glucagon response to hypoglycaemia in 24 people with type 1 diabetes to ascertain whether tight blood glucose control over a period of time improves this response. The investigators aim to achieve good blood glucose control using new generation Automated Insulin Delivery systems (AIDs). This system is made of: an insulin pump, a continuous glucose monitor (CGM) and an algorithm that allows adjustment of insulin delivery based on the blood glucose readings from the CGM. This is the most up to date technology that there is in the management of type 1 diabetes. However, people using this technology often still have problems with high blood glucose after eating. To ensure a very good blood glucose control participants will also follow a low carbohydrate diet to prevent this blood glucose rise after meals.

The Glucagon response to low blood glucose will be measured at zero and eight months using the hyperinsulinaemic hypoglycaemic clamp technique.

DETAILED DESCRIPTION:
This is a feasibility pilot study involving 24 participants with type 1 diabetes. Participants will be recruited from the local type 1 diabetes clinic and insulin pump waiting list. Each participant will enter the trial for a period of 8 months. The investigators aim to test if maximising time in glycaemic range (blood glucose 3.9-10 mmol/L) will restore the glucagon response to insulin-induced hypoglycaemia.

After signing informed consent participants will be screened for eligibility against the inclusion and exclusion criteria.

Those who are eligible will have an initial 20-day period of baseline blood glucose data collection. This will be achieved using a blinded continuous glucose monitoring (CGM) device. Participants will continue on their pre-trial diabetes care during this period and will be required to monitor their own blood glucose as normal.

The participants will be split into two groups using stratified sampling to match for: age, gender and BMI.

Group 1 will be the control group. Participants in this group will continue on standard diabetes care for the duration of the trial. Participants will be required to undertake two further periods of blinded CGM monitoring at 4 and 8 months.

Group 2 will be the intervention group. Participants in this group will be placed on the automated insulin delivery (AID) system and asked to follow a low carbohydrate diet of 30-40g of carbohydrate per main meal portion. The AID system will consist of: a Tandem t:slim X2 insulin pump with control IQ technology and a Dexcom G6 continuous glucose monitor. After receiving training on the use of the devices these participants will enter a 2 week study run-in period to become accustomed to the devices and so that device settings can be optimised. As a safety measure these participants will be asked to measure blood ketones at least once daily throughout the trial. Study staff will monitor the data from the participants study devices throughout the trial and adjust settings as required to maximise time in glycaemic range.

At the beginning and end of the trial all participants will undergo a hyperinsulinaemic hypoglycaemic clamp study to measure their counterregulatory hormone response to hypoglycaemic. Participants will also undergo cognitive tests and assessment of hypoglycaemic awareness during each clamp study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 1 diabetes with C-peptide levels less than 200pmol/L.
* Type 1 diabetes for 5 years or more.
* HbA1c greater than or equal to 53 mol/mol.
* Normal renal function.
* Normal thyroid function.
* Gold Score 4-7 (indicating impaired awareness of hypoglycaemia)
* Willingness to monitor blood ketones daily.
* Use of freestyle libre device is permitted at study entry and may be continued in participants in group 1

Exclusion Criteria:

* Current use of a non-approved closed loop / AID system or those on a predictive low glucose suspend insulin pump.
* Proliferative retinopathy
* Regular use of real time CGM in the preceding 3 months.
* History of Diabetic ketoacidosis in the preceding 6 months.
* Severe hypoglycaemic episode requiring external assistance in the preceding 6 months.
* Inability to safely use technology used in this study (e.g. impaired vision, memory or dexterity that prevents safe operation of CGM or insulin pump.)
* Inability to support the technology requirements for the study (e.g. unable to upload study device at home)
* History of Haemophilia, Cystic Fibrosis, pancreatic disease or complete pancreatectomy, ischaemic heart disease, epilepsy or hypoglycaemia induced seizure
* History of severe reaction or allergy to adhesive necessary to this study.
* Unable to adhere to study timetable.
* Unable to give informed consent.
* Pregnancy. We will perform a pregnancy test on all eligible participants at baseline.
* Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas. These may lower insulin requirements and predispose to diabetic ketoacidosis.
* Concurrent use of medication that may affect blood glucose such as SSRIs
* A condition, which in the opinion of the investigator, would put the patient or study at risk
* HbA1c greater than or equal to 75 mmol/mol

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2025-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shareen Forbes, MBChB, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Edinburgh Royal Infirmary/University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baxter F, Baillie N, Forbes S. Study protocol: a randomised controlled proof-of-concept real-world study - does maximising time in range using hybrid closed loop insulin delivery and a low carbohydrate diet restore the glucagon response to hypoglycaemia in adults with type 1 diabetes? BMJ Open. 2022 Dec 20;12(12):e054958. doi: 10.1136/bmjopen-2021-054958. PMID 36600427

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - Standard Care: Standard diabetes care. They will undergo 3 periods of blinded continuous glucose monitoring (CGM) lasting 20-days at: baseline, 4 and 8 months. Participants in this group will undergo a hyperinsulinaemic hypoglycaemic clamp study at baseline and 8 months and complete quality of life and diabetes treatment questionnaires.
  Stepped hyperinsulinaemic-hypoglycaemic clamp study: Participants will commence a primed insulin infusion at 60mU/m2/min along with a variable rate 20% glucose infusion. Blood glucose monitored (BG) every 5 minutes. The glucose infusion will be altered to achieve BG plateaus of: 5, 3 and 2.5mmol/l. Each lasting 40 minutes. During each plateau blood samples will be taken 3 times for: glucagon, cortisol, adrenaline, noradrenaline, D2 glucose and D5 glycerol. On 2 occasions participants will complete the Edinburgh hypoglycaemia scale and cognitive tests: trail making test, digit span test, digit symbol substitution test and four choice reaction time test. At the end of the clamp study the insulin infusion will be stopped.
  Blinded CGM: Allows data on BG to be collected without values altering behaviour. Participants continue to monitor their own BG while wearing the device in the blinded mode.
  Stable isotope studies- D2 Glucose and D5 Glycerol: takes place at the same time as the hyperinsulinaemic hypoglycaemic clamp. Participants will receive a priming dose of each stable isotope followed by a continuous infusion for the remainder of the clamp study.
- Group 2- Automated Insulin Delivery and Low Carbohydrate Diet: Automated insulin delivery system: Tandem t:slim x2 insulin pump with Control IQ and Dexcom G6 continuous glucose monitor (CGM). They will be asked to follow a low-carbohydrate diet (30-40g of carbs/meal). Baseline 20-day period of blinded CGM. Participants in this group will undergo a stepped hypoglycaemic clamp study at baseline and 8 months and complete quality of life and diabetes treatment questionnaires.
  Stepped hypoglycaemic clamp study: Participants commence a primed insulin infusion (rate 60mU/m2/min) and a variable rate 20% glucose infusion. Blood glucose (BG) monitored every 5 minutes. Glucose infusion will be altered to achieve BG plateaus of: 5, 3 and 2.5mmol/l. Each lasting 40 minutes. During each plateau blood samples will be taken 3 times for: glucagon, cortisol, adrenaline, noradrenaline, D2 glucose and D5 glycerol. Twice during each plateau participants complete the Edinburgh hypoglycaemia scale and cognitive tests: trail making test, digit span test, digit symbol substitution test and four choice reaction time test.
  Insulin pump: Insulin pump with a built-in algorithm automatic insulin adjustment.
  CGM: CGM sends data to the insulin pump to allow automatic insulin adjustment.
  Low carbohydrate diet: 30-40g of carbs/meal.
  Blinded CGM: data on BG collected without values altering behaviour.
  Stable isotope studies- D2 Glucose and D5 Glycerol: These studies will take place at the same time as the hypoglycaemic clamp.
Period: Overall Study
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Started | 8 | 11
Completed | 5 | 11
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (11.3) | 42.9 (9.5) | 39.95 (10.63)
Sex/Gender, Customized [Number; unit: participants]
  Female | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 11 | 19
Age Diagnosed (Years) [Median (Inter-Quartile Range); unit: Years] | 7 [3 to 32] | 20 [7 to 31] | 16.5 [4.75 to 31.25]
Time since diagnosis (Years) [Median (Inter-Quartile Range); unit: Years] | 19.2 [14 to 28.1] | 25.5 [11 to 32] | 24.67 [12.5 to 31.29]
HbA1c [Median (Inter-Quartile Range); unit: mmol/mol] | 63 [63 to 64.8] | 61 [57 to 68] | 63 [58 to 65]
Weight [Mean (Standard Deviation); unit: Kg] | 84.5 (11.9) | 77.33 (7.8) | 80.35 (10.14)
BMI [Mean (Standard Deviation); unit: kg^m2] | 29.34 (4.1) | 26.18 (2.99) | 27.51 (3.76)
Insulin Pump User [Number; unit: participants] | 4 | 3 | 7
Time in range (3.9-10 mmol/L) [Mean (Standard Deviation); unit: Percentage time spent 3.9-10 mmol/L] | 49.05 (12.47) | 53.55 (14.48) | 50.39 (13.83)
Time <3.9 mmol/L [Median (Inter-Quartile Range); unit: Percentage] | 0.71 [0.44 to 1.78] | 0.65 [0.39 to 3.28] | 0.71 [0.39 to 2.27]
Time <3.0 mmol/L [Median (Inter-Quartile Range); unit: Percentage] | 0.12 [0.00 to 0.19] | 0.13 [0.03 to 0.52] | 0.13 [0.03 to 0.32]
Time >10 mmol/L [Mean (Standard Deviation); unit: Percentage] | 25.12 (11.73) | 33.64 (12.42) | 30.05 (12.57)
Time >13.9 mmol/L [Mean (Standard Deviation); unit: Percentage] | 21.7 (8.77) | 15.25 (13.75) | 17.97 (12.07)
CV Glucose [Mean (Standard Deviation); unit: Percentage] | 38.24 (6.8) | 35.06 (4.94) | 36.4 (5.85)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Plasma Glucagon Levels (Pmol/L) Measured During Normoglycaemic and Hypoglycaemia
Description: The delta glucagon concentration (pmol/L) from plateau 1 (normoglycaemia- 5.0 mmol/L) to plateau 3 (hypoglycaemia- 2.5 mmol/L). The physiological response in health would be for an increase in glucagon secretion from normo- to hypoglycaemia.
Time Frame: Clamp 1 at baseline and clamp 2 at 8 months
Population: Three participants withdrew from group 1 after the 1st clamp study visit. They were excluded from the study analysis.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
pmol/L
  Delta Clamp 1 (P3-P1) | 1.34 [0.46 to 4.52] | 1.68 [0.96 to 3.35]
  Delta Clamp 2 (P3-P1) | 2.26 [0.52 to 3.64] | 0.31 [0.00 to 1.53]
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time in Glycaemic Range (3.9-10mmol/L)
Description: Percentage time spent in target glycaemic range.
Time Frame: Baseline (study entry), midpoint at 4 months and endpoint at 8 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Percentage
  Baseline | 51.46 (13.63) | 53.55 (14.48)
  Midpoint | 44.26 (11.5) | 78.01 (6.32)
  Endpoint | 39.64 (20.15) | 76.85 (9.61)
Statistical Analysis 1: Comparison: Group 1 - Standard Care vs Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.37, ANOVA
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p < 0.0001, ANOVA

3. Secondary Outcome: Time Spent Below the Target Glycaemic Range (<3.9mmol/L)
Description: Percentage of time spent below the target glycaemic range
Time Frame: Baseline (study entry), midpoint at 4 months and endpoint at 8 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Percentage
  Baseline | 1.02 (0.62) | 2.13 (3.17)
  Midpoint | 2.25 (3.50) | 0.94 (0.55)
  Endpoint | 2.18 (3.85) | 0.74 (0.57)
Statistical Analysis 1: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.20, ANOVA
Statistical Analysis 2: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.95, ANOVA

4. Secondary Outcome: Time Spent Above the Target Glycaemic Range (>10mmol/L)
Description: Percentage of time spent above the target glycaemic range
Time Frame: Baseline (study entry), midpoint at 4 months and endpoint at 8 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Percentage
  Baseline | 21.94 (13.93) | 33.64 (12.42)
  Midpoint | 21.67 (13.55) | 18.93 (4.66)
  Endpoint | 23.42 (17.23) | 19.06 (5.87)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.58, ANOVA
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.01, ANOVA

5. Secondary Outcome: The Change in Plasma Cortisol (ng/mL) Levels Measured During Normoglycaemic and Hypoglycaemia
Description: Delta cortisol from P1 (5.0 mmol/L) to P3 (2.5 mmol/L)
Time Frame: Clamp 1 at baseline and clamp 2 at 8 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
ng/mL
  Delta P3-P1 Clamp 1 | 146 (126) | 72.52 (91.48)
  Delta P3-P1 Clamp 2 | 195.2 (115.9) | 11.31 (37.14)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: The Change in Plasma Adrenaline (pg/mL) Levels Measured During Normoglycaemic and Hypoglycaemia
Description: Delta adrenaline from plateau 1 (5mmol/L) to plateau 3 (2.5 mmol/L)
Time Frame: Clamp 1 at baseline and clamp 2 at 8 months
Measure: Median (Inter-Quartile Range); unit: Delta pg/mL
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Delta pg/mL
  Clamp 1 | 260 [78.5 to 499] | 187 [27.25 to 658.5]
  Clamp 2 | 413 [267.5 to 524.5] | 252.5 [172.8 to 696.5]
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: The Change in Plasma Noradrenaline (pg/mL) Levels Measured During Normoglycaemic and Hypoglycaemia
Description: The change in noradrenaline concentration from plateau 1 (5 mmol/L) to plateau 3 (2.5 mmol/L).
Time Frame: Clamp 1 at baseline and clamp 2 at 8 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
pg/mL
  Delta noradrenaline (P3-P1) Clamp 1 | 49 [-132 to 225] | -10.56 [-50.25 to 38.75]
  Delta noradrenaline (P3-P1) Clamp 2 | -43 [-133 to 56] | 90.5 [3.75 to 172.3]
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Endogenous Glucose Production
Description: The change in the glucose rate of appearance from plateau 1 (5mmol/L) to plateau 3 (2.5 mmol/L)
Time Frame: Clamp 1 at baseline and clamp 2 at 8 months
Measure: Mean (Standard Deviation); unit: mg/kg/minute
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
mg/kg/minute
  Delta glucose rate of appearance P3-P1 Clamp 1 | -0.16 (0.21) | -0.12 (0.16)
  Delta glucose rate of appearance P3-P1 Clamp 2 | -0.22 (0.16) | -0.8 (0.16)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.88, t-test, 2 sided

9. Secondary Outcome: HbA1c
Description: Delta HbA1c from baseline to study endpoint.
Time Frame: Baseline (study entry) endpoint (8 months)
Measure: Median (Inter-Quartile Range); unit: mmol/mol
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
mmol/mol | 0 [-4.5 to 4] | -12 [-18 to -4]
Statistical Analysis 1: Comparison: Group 1 - Standard Care vs Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.0094, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Quality of Life at Trial Entry and End.
Description: Measured using the EQ5D-5L- -VAS. Number on scale of 0-100 to assess wellbeing on that day. 100 being the most well.
Time Frame: Baseline (study entry) endpoint (8 months)
Measure: Mean (Standard Deviation); unit: Number
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Number
  Baseline | 81 (6.52) | 79.36 (12.33)
  Endpoint | 82 (11.51) | 80.27 (9.96)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.82, t-test, 2 sided

11. Secondary Outcome: Change in Emotional Distress Related to Diabetes at Trial Entry and End.
Description: Diabetes Distress Scale (DDS-1)- a 28-item self-reporting scale. Each item can be scored from 1 (not a problem) to 6 (a very serious problem). This questionnaire will be completed at study entry and study end. Data presented is the DDS total score.
Time Frame: Baseline (study entry) endpoint (8 months)
Measure: Mean (Standard Deviation); unit: Numerical score
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Numerical score
  Baseline | 2.18 (0.64) | 2.2 (1.15)
  Endpoint | 1.96 (0.66) | 1.58 (0.49)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Fear of Hypoglycaemic
Description: Measured using the Hypoglycaemia Fear Survey (HFS)- this survey consists of two subscales- Baseline (study entry) endpoint (8 months) Behaviour and Worry. There are 28 items in the survey that the participant ranks from Never (0) to Almost Always (4). Higher scores indicate fear of hypoglycaemia. In the Behaviour subscale the lowest possible score in 0 and the highest possible score is 60. In the Worry subscale the lowest possible score is 0 and the highest is 72.
  Participants will complete this questionnaire at study entry and study end.
Time Frame: Baseline (study entry) endpoint (8 months)
Measure: Mean (Standard Deviation); unit: Numerical score
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Numerical score
  Behaviour Scale Baseline | 22 (4.24) | 20.55 (4.03)
  Behaviour Scale Endpoint | 19.2 (8.11) | 18.82 (4.79)
  Worry scale Baseline | 24 (9.34) | 24.25 (15.85)
  Worry Scale Endpoint | 21.4 (15.39) | 12.88 (9.78)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Behaviour subscale; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Standard Care; Worry subscale; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Behaviour subscale; Test type: Superiority; p = 0.35, t-test, 2 sided
Statistical Analysis 4: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Worry subscale; Test type: Superiority; p = 0.09, t-test, 2 sided

13. Secondary Outcome: Change in Confidence of Managing Hypoglycaemia
Description: Measured using the Hypoglycaemic Confidence Scale- this is a 9 item scale. The participant rates each item from Not Confident at All to Very Confident. Participants will complete this questionnaire at study entry and study end. Higher scores mean more confidence. 'Not confident' at lower end of scale scored as 1 and 'very confident' at top of the scale scored as 4. Min score is 9 and max score is 36.
Time Frame: Baseline (study entry) endpoint (8 months)
Measure: Mean (Standard Deviation); unit: Numerical score
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Numerical score
  Baseline | 27.2 (5.17) | 27.64 (7.63)
  Endpoint | 29.2 (5.31) | 31.27 (3.9)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.09, t-test, 2 sided

14. Secondary Outcome: Hypoglycaemia Awareness
Description: Measured during each clamp study using the Edinburgh Hypoglycaemic Scale- this is a 17 item scale of symptoms of hypoglycaemia. The participant ranks on a scale from Not at all (1) to A Great Deal (7) whether they are experiencing each symptom at the time of the questionnaire being completed. Higher scores mean more hypoglycaemia symptoms. The lowest possible score is 0 and the highest possible score is 119.
Time Frame: Clamp 1 - study entry, clamp 2 - 8 months
Measure: Median (Inter-Quartile Range); unit: Numerical score
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Numerical score
  Clamp 1 Plateau 1 | 24 [22.5 to 31.5] | 27 [18 to 32]
  Clamp 1 Plateau 2 | 35 [29.5 to 60.5] | 25 [19 to 50]
  Clamp 1 Plateau 3 | 39.64 [30.5 to 62.5] | 34 [24 to 64]
  Clamp 2 Plateau 1 | 34 [23.5 to 36] | 28 [22 to 36]
  Clamp 2 Plateau 2 | 34 [27 to 64.5] | 29 [24 to 60]
  Clamp 2 Plateau 3 | 46 [29.5 to 71] | 47 [26 to 76]
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.77, ANOVA — Column factor p-value
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.37, ANOVA

15. Secondary Outcome: Trial Making Test
Description: Measured during each plateau in a stepped hypoglycaemic clamp study at study entry and study end. Delta score plateau 1 (5 mmol/L) to plateau 3 (2.5 mmol/L) compared between clamp studies. Participants are timed completing the test. Higher scores indicate a longer time to complete the test.
Time Frame: Clamp 1- study entry, clamp 2 - 8 months
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Minutes
  Trail making A delta clamp 1 | -3.05 [-4.55 to 0.4] | 0.00 [-12.0 to 1.50]
  Trail making A delta clamp 2 | -2.6 [-4.55 to 0.05] | -1.9 [-7.2 to 2.4]
  Trail making B delta clamp 1 | 11.5 [-10.35 to 22.8] | -7.8 [-10.0 to 1.0]
  Trail making B delta clamp 2 | 0.7 [-2.98 to 5.5] | -5.6 [-23.9 to -0.9]
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Trail making A delta clamp 1 compared to clamp 2; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Standard Care; Trail Making B delta clamp 1 compared to clamp 2; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Trail making A delta clamp 1 compared to clamp 2; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Trail making B delta clamp 1 compared to clamp 2; Test type: Superiority; p = 0.49, t-test, 2 sided

16. Secondary Outcome: Digit Span Test
Description: Measured during each plateau in a stepped hypoglycaemic clamp study at study entry and study end. Difference in change in score from plateau 1 (5mmol/L) to plateau 3 (2.5 mmol/L) compared between clamp studies. Lower scores mean more errors. Forwards- participant repeats the numbers as read. Backwards- the participant repeats the numbers backwards.
Time Frame: Clamp 1- study entry, clamp 2 - 8 months
Measure: Median (Inter-Quartile Range); unit: Correct responses
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Correct responses
  Digit span forwards clamp1 | -1 [-2 to 0] | -1 [-1 to 1]
  Digit span forwards clamp 2 | 0 [-1.5 to 1.5] | 0 [-1 to 0]
  Digit span backwards clamp 1 | 0 [-1 to 0] | 0 [-1 to 0]
  Digit span backwards clamp 2 | 0 [-1 to 2] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Digit span forwards; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Standard Care; Digit span backwards; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Digit span forwards; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Digit Symbol Substitution Test
Description: Measured during each plateau in a stepped hypoglycaemic clamp study at study entry and study end. Difference in score between plateau 1 (5.0 mmol/L) and plateau 3 (2.5 mmol/L) compared between clamp studies. Given 90 seconds to complete as many items as possible. Higher scores mean more items completed in the allotted time.
Time Frame: Clamp 1- study entry, clamp 2 - 8 months
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Correct responses
  Delta score clamp 1 | -4.4 (5.4) | 0.82 (6.56)
  Delta score clamp 2 | -6.6 (13.7) | -4.0 (7.1)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.06, t-test, 2 sided

18. Secondary Outcome: Four Choice Reaction Time Test
Description: Measured during each plateau in a stepped hypoglycaemic clamp study at study entry and study end. Difference in score between plateau 1 (5.0mmol/L) and plateau 3 (2.5 mmol/L) compared between clamp studies. Higher scores mean more time taken to complete the task.
Time Frame: Clamp 1- study entry, clamp 2 - 8 months
Measure: Mean (Standard Deviation); unit: Time (ms)
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
Number analyzed (Participants) | 5 | 11
Time (ms)
  Clamp 1 | 15.4 (7.4) | 38.45 (63.21)
  Clamp 2 | 52.9 (20.43) | 57.78 (60.63)
Statistical Analysis 1: Comparison: Group 1 - Standard Care; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 2- Automated Insulin Delivery and Low Carbohydrate Diet; Test type: Superiority; p = 0.27, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From recruitment of participant to study completion (8 months per participants).
Arm/Group | Group 1 - Standard Care | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/11
Other Adverse Events (participants affected / at risk) | 0/5 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Standard Care (N=5) | Group 2- Automated Insulin Delivery and Low Carbohydrate Diet (N=11)
Proliferative retinopathy (Eye disorders) | 0 (0) | 1 (1) — 3 month eye screening one participant HCL group was diagnosed with proliferative retinopathy in their left eye (R1 to R4). They were referred to ophthalmology. Repeat screening by ophthalmology showed R1 in both eyes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT04614168/Prot_SAP_001.pdf